CLINICAL TRIAL: NCT01816230
Title: Allogeneic Stem Cell Transplantation of NiCord®, Umbilical Cord Blood-derived Ex Vivo Expanded Stem and Progenitor Cells, in Adolescent and Adult Patients With Hematological Malignancies
Brief Title: Transplantation of NiCord®, Umbilical Cord Blood-derived Ex Vivo Expanded Cells, in Patients With HM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#03.01.020
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hematological Malignancies; Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NiCord® (Experimental): NiCord® is a stem/progenitor cell based product composed of ex vivo expanded allogeneic UCB cells.
  Interventions: Drug: NiCord®

INTERVENTIONS:
Drug: NiCord®

SUMMARY:
A Study Evaluating the Safety and Efficacy of Transplantation of a single cord blood unit (CBU) of NiCord®, umbilical cord blood-derived Ex Vivo Expanded Stem and Progenitor Cells in Patients with Hematological Malignancies.

DETAILED DESCRIPTION:
Umbilical cord blood (UCB) is an alternative stem cell source for hematopoietic stem cell transplantations (HSCT) and can be used for the treatment of various life-threatening diseases, such as hematological malignancies or genetic blood disorders, in such cases where a matched related stem cell donor is not available. However, the major drawback of using this valuable stem cells source is the limited cell dose in a single cord blood unit (CBU), which was shown to be associated with inadequate hematopoietic reconstitution and high risk of transplant-related mortality. To improve outcomes and extend applicability of UCB transplantation, one potential solution is ex vivo expansion of UCB-derived stem and progenitor cells. NiCord® is a stem/progenitor cell based product composed of ex vivo expanded allogeneic UCB cells. NiCord® is based on a novel technology for the ex vivo cell expansion of cord blood derived hematopoietic progenitor cells. By increasing the number of the short and long-term reconstitution progenitor cells transplanted, NiCord® has the potential to enable the broader application of UCB transplantation, and improve the clinical outcomes of UCB transplantation.

The study is designed as a multi center, single arm study, evaluating the safety and efficacy of the transplantation of NiCord® to patients with hematological malignancies following myeloablative therapy.

Total study duration is approximately 400 days from the signing of informed consent to the last visit one year following transplantation

The overall study objective is to evaluate the safety and efficacy of NiCord®: single ex-vivo expanded cord blood unit transplantation in patients with hematological malignancies following myeloablative therapy as follows:

The main study objectives are to assess the cumulative incidence of patients with NiCord®-derived neutrophil engraftment at 42 days following transplantation and to assess the incidence of secondary graft failure at 180 days following transplantation of NiCord® Ten evaluable patients recruited for the study should be 12-65 years of age, up to a maximum of 15 treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Applicable disease and eligible for myeloablative SCT
* Patients must have two partially HLA-matched CBUs
* Back-up stem cell source
* Adequate Karnofsky Performance score or Lansky Play-Performance scale
* Sufficient physiological reserves
* Signed written informed consent

Exclusion Criteria:

* HLA-matched donor able to donate
* Prior allogeneic HSCT
* Other active malignancy
* Active or uncontrolled infection
* Active/symptoms of central nervous system (CNS) disease
* Pregnancy or lactation

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke University
Locations (15):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Steven and Alexandra Cohen Children's Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt, Nashville, Tennessee
- Italy (2):
  - Children Hospital Gaslini Scientific Institute, Genoa
  - University of Turin, Turin
- University Medical Center Utrecht, Utrecht, Netherlands
- Singapore (2):
  - National University Cancer Institute, Singapore
  - Singapore General Hospital, Singapore
- Spain (2):
  - University Hospital Vall d´Hebron, Barcelona
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Derived] Horwitz ME, Wease S, Blackwell B, Valcarcel D, Frassoni F, Boelens JJ, Nierkens S, Jagasia M, Wagner JE, Kuball J, Koh LP, Majhail NS, Stiff PJ, Hanna R, Hwang WYK, Kurtzberg J, Cilloni D, Freedman LS, Montesinos P, Sanz G. Phase I/II Study of Stem-Cell Transplantation Using a Single Cord Blood Unit Expanded Ex Vivo With Nicotinamide. J Clin Oncol. 2019 Feb 10;37(5):367-374. doi: 10.1200/JCO.18.00053. Epub 2018 Dec 4. PMID 30523748

RESULTS

PARTICIPANT FLOW:
Groups:
- NiCord®: NiCord® is a stem/progenitor cell based product composed of ex vivo expanded allogeneic UCB cells.
  NiCord®
Period: Overall Study
Arm/Group | NiCord®
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- NiCord®: NiCord® is a stem/progenitor cell based product composed of ex vivo expanded allogeneic umbilical cord blood (UCB) cells.
  NiCord®
Arm/Group | NiCord®
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: Years] | 44 [13 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Primary diagnosis [Count of Participants; unit: Participants]
  Acute lymphoblastic leukemia (ALL) | 9
  Adult acute myeloid leukemia (AML) | 17
  Myelodysplastic syndromes (MDS) | 7
  non-Hodgkins Lymphoma | 0
  Hodgkins Disease | 1
  Chronic myeloid leukemia (CML) | 2
Adjusted disease risk index [Count of Participants; unit: Participants]
  Low | 8
  Intermediate | 15
  High | 13

OUTCOME MEASURES:

1. Primary Outcome: Engraftment
Description: Assess the cumulative incidence of patients with NiCord®-derived neutrophil engraftment at 42 days following transplantation.
Time Frame: 42 days
Measure: Number; unit: percentage of patients
Arm/Group | NiCord®
Number analyzed (Participants) | 36
percentage of patients | 94

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | NiCord®
All-Cause Mortality (participants affected / at risk) | 16/36
Serious Adverse Events (participants affected / at risk) | 34/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NiCord® (N=36)
Infection (Infections and infestations) | 17
GvHD (Immune system disorders) | 11
Hematologic Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NiCord® (N=36)
Decreased appetite (Metabolism and nutrition disorders) | 9
Hypertension (Vascular disorders) | 13
Leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 6
GvHD (Immune system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT01816230/Prot_SAP_000.pdf